CLINICAL TRIAL: NCT05818085
Title: A Multicenter, Randomized, Double-blind, Controlled, Phase 2b/3 Study to Assess the Efficacy and Safety of ABP-671 in Participants With Gout
Brief Title: Phase 2b/3 Study to Assess ABP-671 a Novel URAT1 Inhibitor in Participants With Gout
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-671-301
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABP-671 (Experimental)
  Interventions: Drug: ABP-671
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ABP-671 — Low, medium or high dose (Part 1); Selected dose(s) (Part 2)
  Arms: ABP-671
Drug: Allopurinol — Standard of care according to American College of Rheumatology (ACR) guideline for the management of gout
  Arms: Allopurinol
Other: Placebo — ABP-671 matching placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, Phase 2b/3 study to evaluate the efficacy and safety of ABP-671. Part 1 of the study will compare the efficacy and safety of different doses and regimens of ABP-671 with placebo and allopurinol. Part 2 of the study will compare the dosing regimen(s) of ABP-671 selected from Part 1 with placebo in participants who have not been enrolled for Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥19 and <70 years of age at the time of informed consent.
* A body mass index (BMI) of ≥18 kg/m2 to ≤40 kg/m2.
* Diagnosis of gout per American College of Rheumatology/European Alliance of Associations for Rheumatology 2015 Gout Classification Criteria and must meet the criteria as follows:

  * At Screening, participants with gout on ULT (including allopurinol) must be willing to discontinue ULT.
  * At Screening, participants with gout who are not currently treated with any UA lowering therapy must have an sUA ≥7.5 mg/dL (≥0.450 mmol/L).
* At the confirmatory sUA visit, all participants must have an sUA ≥7.0 mg/dL (≥0.420 mmol/L).
* Women of childbearing potential (WOCBP) must be surgically sterile (eg, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or willing to use acceptable and highly effective double contraception from Screening until at least 30 days after the last dose of the study drug. Double contraception is defined as a condom AND one other form of the following:

  * Established hormonal contraception (with approved oral contraceptive pills, long-acting implantable hormones, injectable hormones);
  * A vaginal ring or an intrauterine device OR
  * Documented evidence of surgical sterilization at least 6 months prior to Screening (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is the sole partner). The absence of records will not exclude screening the participant; if medical records cannot be obtained, serum pregnancy testing will be conducted to confirm the participant is not pregnant.

Note: Women not of childbearing potential must be postmenopausal for ≥12 months. Postmenopausal status will be confirmed through follicle stimulating hormone (FSH) concentration testing.

-Men must be surgically sterile (>30 days since vasectomy), abstinent, or if engaged in sexual relations with a female partner of childbearing potential, the participant must use an acceptable form of contraception from Screening until at least 30 days after the last dose of the study drug. Acceptable methods of contraception include the use of condoms in addition to the use of an effective contraceptive for the female partner that includes approved oral contraceptive pills, long-acting implantable hormones, injectable hormones, a vaginal ring, or an intrauterine device. Participants who practice abstinence (abstinence from penile-vaginal intercourse) are eligible when this is in line with their preferred and usual lifestyle. In addition, men must not donate sperm for at least 30 days after the last dose of the study drug.

Exclusion Criteria:

* History of rheumatoid arthritis or other autoimmune disease.
* Clinically significant hepatic, cardiovascular, renal, neoplastic, psychiatric, or hematological disorders such as polycythemia vera, sickle cell disease, or myelodysplastic disorder.
* Positive test result for HIV, hepatitis B surface antigen, or hepatitis C virus antibody. Active hepatitis C virus infection is defined as a participant with a positive hepatitis C antibody and detectable hepatitis C viral load RNA.
* Participants who, in the opinion of the Investigator, have a high genetic risk of allopurinol hypersensitivity syndrome unless they have been found to be negative for Human leukocyte antigen (HLA)-B*5801, either clinically by prior exposure to allopurinol or by laboratory evaluation.
* Liver function tests >2x the laboratory upper limit of normal (ULN) range of aspartate aminotransferase, alkaline phosphatase, or alanine aminotransferase; total bilirubin >1.5x ULN at Screening.
* Inadequate renal function with serum creatinine >1.5 mg/dL (>0.133 mmol/L) or estimated glomerular filtration rate (eGFR) < 60 mL/min/m2 (by the 2021 Chronic Kidney Disease Epidemiology Collaboration creatinine-based eGFR equation).
* History of malignancy within the previous 5 years; with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia, or treated in situ grade 1 cervical cancer.
* History within the last 12 months of unstable angina, New York Heart Association functional class III or IV heart failure, myocardial infarction, stroke, venous thromboembolism, or a history of percutaneous coronary intervention.
* Uncontrolled hypertension (systolic BP ≥160 mmHg and/or diastolic BP ≥90 mmHg). If BP is controlled while taking antihypertensive medication, the participant must be on stable dose for previous 2 months.
* Active liver disease or impaired hepatic function as assessed by liver function tests.
* Received any investigational therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening.
* Any other medical or psychological condition, that, in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the participant, interfere with the participant's ability to comply with the protocol requirements to complete the study, or potentially compromise the results or interpretation of the study.
* Pregnant, breastfeeding, or planning a pregnancy during the study or ≤30 days after the last dose of the study drug.
* Intolerant or unwilling to take colchicine or naproxen.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve serum uric acid (sUA) levels <6.0 mg/dL (<0.360 mmol/L) | Week 28

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and Tolerability) | Week 28
  Incidence of treatment-emergent adverse events (TEAEs), including AEs of special interest (AESIs), serious AEs (SAEs), and AEs leading to study treatment discontinuation
Proportion of participants who achieve sUA levels <5.0 mg/dL (<0.300 mmol/L) | Week 28

CONTACTS AND LOCATIONS:
Locations (56):
- United States (35):
  - Alliance for Multispecialty Research, Tempe, Arizona
  - Tucson Neuroscience Research, LLC, Tuscon, Arizona
  - Anaheim Clinical Trials (Cenexel ACT), Anaheim, California
  - Center for Clinical Trials of Sacramento, Sacramento, California
  - Access Research Institute, Brooksville, Florida
  - Nature Coast Clinical Reasearch, Crystal River, Florida
  - JY Research Institute Inc., Cutler Bay, Florida
  - Accel Clinical Research Site, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Accel Research Sites Network - St. Pete-Largo Clinical Research Unit, Largo, Florida
  - A & D Doctor Center, Miami, Florida
  - Bioclinical Research Alliance, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Century Research LLC, Miami, Florida
  - ITB Research, Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - New Horizons Research, Palmetto Bay, Florida
  - Advanced Clinical Research of Atlanta, Atlanta, Georgia
  - Centricity Research, Columbus, Georgia
  - Alliance for Multispecialty Research, LLC., Newton, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - AMR, New Orleans, Louisiana
  - Annapolis Internal Medicine/CCT Research, Annapolis, Maryland
  - DelRicht Research of Gulfport, Gulfport, Mississippi
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Santa Rosa Medical Center, Las Vegas, Nevada
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - OnSite Clinical Solutions, Salisbury, North Carolina
  - DelRicht Research, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Medical Care/CCT, Elizabethton, Tennessee
  - PanAmerican Clinical Research, LLC, Brownsville, Texas
  - Quality Research Inc., San Antonio, Texas
  - Centricity Research, Suffolk, Virginia
- Australia (6):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research Sydney, Botany, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - A R Houston Medical Pty Ltd, Kippa-Ring, Queensland
  - Emeritus Research Melbourne, Camberwell, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg, Victoria
- Georgia (6):
  - New Hospitals, Tbilisi
  - Evex Hospitals Caraps Medline, Tbilisi
  - Aversi Clini, Tbilisi
  - The First Medical Center, Tbilisi
  - Academician Vakhtang Bochorishvili Clinic, Tbilisi
  - Innova, Tbilisi
- Guatemala (4):
  - Clinical Research Center (CRC), Guatemala City
  - Clínica Médica Especializada en Medicina Interna y Reumatología (CREER), Guatemala City
  - Clínica Médica Especializada en Medicina Interna y Reumatología, Guatemala City
  - Clínica Médica Especializada en Medicina Interna, Guatemala City
- Taiwan (5):
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Memorial Hospital CGMH, Kaohsiung City
  - Chung Shan Medical Univ. Hospital, Taichung
  - Cheng-Shin General Hospital, Taipei
  - Chang Gung Memorial Hospital LinKou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No